CLINICAL TRIAL: NCT07363187
Title: Evaluation of Microvascular Changes by Nailfold Capillaroscopy and Serum ADMA, Von Willebrand Factor, Hs-CRP, and D-dimer Levels in Healthcare Workers Exposed to Chronic Low-Dose Ionizing Radiation
Brief Title: Nailfold Capillaroscopy and Endothelial Biomarkers in Healthcare Workers Exposed to Chronic Low-Dose Ionizing Radiation
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Banu Yildiran, Dermatology Resident Physician, Istanbul Training and Research Hospital
Other Study IDs: SBU-IEAH-EC274
Record Dates: First submitted 2026-01-07; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Microvascular Dysfunction; Endothelial Dysfunction; Occupational Radiation Exposure
Keywords: Nailfold capillaroscopy; Microvascular changes; Low-dose ionizing radiation; Occupational radiation exposure; Healthcare workers; Endothelial dysfunction; Inflammation biomarkers; D-dimer; High-sensitivity C-reactive protein; Asymmetric dimethylarginine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Venous blood samples will be collected from all participants. Serum samples will be obtained after centrifugation. Von Willebrand factor (vWF) and D-dimer levels will be measured using routine hospital biochemistry laboratory methods. Serum samples for the measurement of asymmetric dimethylarginine (ADMA) and high-sensitivity C-reactive protein (hs-CRP) will be aliquoted and stored at -80°C until analysis by ELISA methods. No DNA extraction or genetic analyses will be performed, and all samples will be used exclusively for the purposes defined in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radiation-Exposed Healthcare Workers: Healthcare workers with chronic occupational exposure to low-dose ionizing radiation as part of their routine professional activities in medical departments where radiation is used.
- Non-Exposed Control Group: Healthcare workers without occupational exposure to ionizing radiation, working in departments where radiation-based procedures are not used.

SUMMARY:
Chronic occupational exposure to low-dose ionizing radiation may lead to subclinical endothelial dysfunction and early microvascular alterations in healthcare workers. Nailfold capillaroscopy is a non-invasive method that allows direct visualization of microcirculatory changes. This observational study aims to evaluate microvascular alterations using nailfold capillaroscopy and to assess their association with serum endothelial and inflammatory biomarkers, including asymmetric dimethylarginine (ADMA), von Willebrand factor (vWF), high-sensitivity C-reactive protein (hs-CRP), and D-dimer levels. Healthcare workers with chronic low-dose radiation exposure will be compared with non-exposed controls. The study seeks to improve understanding of early vascular effects of occupational radiation exposure.

DETAILED DESCRIPTION:
Chronic occupational exposure to low-dose ionizing radiation may result in subclinical endothelial dysfunction and early microvascular alterations, even in the absence of overt clinical disease. Healthcare workers employed in medical departments where ionizing radiation is routinely used are exposed to cumulative radiation over time. Identifying early vascular changes in this population is important for understanding potential long-term cardiovascular risks associated with occupational radiation exposure.

Nailfold capillaroscopy is a non-invasive and reproducible imaging technique that enables direct visualization of the microcirculation and allows detailed assessment of capillary density, morphology, and structural abnormalities. Additionally, circulating endothelial and inflammatory biomarkers such as asymmetric dimethylarginine (ADMA), von Willebrand factor (vWF), high-sensitivity C-reactive protein (hs-CRP), and D-dimer may reflect endothelial dysfunction, inflammation, and prothrombotic activity at a subclinical level.

This single-center, observational, cross-sectional study will include healthcare workers with chronic occupational exposure to low-dose ionizing radiation and a control group of healthcare workers without radiation exposure from the same institution. Demographic characteristics, occupational exposure duration, and work-related radiation exposure history will be recorded for all participants.

All participants will undergo nailfold capillaroscopy evaluation using standardized assessment criteria, including capillary density, tortuosity, dilatation, dystrophic changes, avascular areas, microhemorrhages, neoangiogenesis, and subpapillary plexus visibility. Venous blood samples will be collected to measure serum ADMA, vWF, hs-CRP, and D-dimer levels using routine laboratory methods and enzyme-linked immunosorbent assay techniques, as appropriate.

The primary objective of this study is to identify microvascular changes detected by nailfold capillaroscopy in healthcare workers exposed to chronic low-dose ionizing radiation. Secondary objectives include evaluating the association between capillaroscopic findings, serum biomarkers, and occupational radiation exposure characteristics. The findings of this study may contribute to improved understanding of early vascular effects of chronic occupational radiation exposure and support the use of nailfold capillaroscopy as a practical screening tool in exposed populations.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers aged between 18 and 60 years.
* For the control group: Employment in a healthcare institution with either occupational exposure to low-dose ionizing radiation or no occupational radiation exposure.
* For the exposed group: chronic occupational exposure to ionizing radiation for at least 3 years.
* Willingness and ability to provide written informed consent.
* Ability to comply with study procedures, including nailfold capillaroscopy and blood sample collection.

Exclusion Criteria:

* History of cardiovascular disease, cerebrovascular disease, or peripheral vascular disease.
* Presence of systemic diseases that may affect microvascular structure or endothelial function, including diabetes mellitus, uncontrolled hypertension, dyslipidemia, or chronic kidney disease.
* Known autoimmune, connective tissue, or systemic inflammatory diseases (e.g., systemic sclerosis, lupus erythematosus, vasculitis).
* Active infection or acute inflammatory condition at the time of enrollment.
* Use of systemic medications that may affect endothelial function or microcirculation within the past 4 weeks, including vasodilators, antihypertensive agents, statins, antiplatelet or anticoagulant drugs.
* Current smoking or history of smoking within the past 6 months.
* Pregnancy or breastfeeding.
* History of malignancy or current cancer treatment.
* Previous finger trauma, surgery, or local conditions affecting the nailfold area that may interfere with capillaroscopic evaluation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of healthcare workers aged 18 to 60 years employed at a tertiary care hospital. The exposed group will include healthcare workers with chronic occupational exposure to low-dose ionizing radiation, while the control group will include healthcare workers without occupational radiation exposure, working in non-radiation-related departments within the same institution. Participants will be recruited on a voluntary basis and will undergo a single study visit including nailfold capillaroscopy, blood sample collection, and completion of demographic and occupational exposure questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Microvascular Changes Assessed by Nailfold Capillaroscopy | Baseline (single assessment at study visit
  Microvascular alterations will be evaluated using nailfold capillaroscopy, including capillary density and morphological abnormalities such as tortuosity, dilatation, elongated capillaries, dystrophic changes, avascular areas, microhemorrhages, neoangiogenesis, and subpapillary plexus visibility. Capillaroscopic findings will be assessed using standardized semi-quantitative scoring criteria

SECONDARY OUTCOMES:
Serum Asymmetric Dimethylarginine (ADMA) Level | Baseline (single assessment at study visit)
  Serum levels of asymmetric dimethylarginine (ADMA) will be measured as a marker of endothelial dysfunction.
Serum von Willebrand Factor (vWF) Level | Baseline (single assessment at study visit)
  Serum von Willebrand factor (vWF) levels will be measured to assess endothelial activation and vascular injury.
Serum High-Sensitivity C-Reactive Protein (hs-CRP) Level | Baseline (single assessment at study visit)
  Serum high-sensitivity C-reactive protein (hs-CRP) levels will be measured as a marker of systemic inflammation.
Serum D-dimer Level | Baseline (single assessment at study visit)
  Serum D-dimer levels will be measured to evaluate prothrombotic activity.
Correlation Between Nailfold Capillaroscopy Scores and Serum Biomarker Levels | Baseline (cross-sectional analysis)
  The correlation between nailfold capillaroscopy findings and serum biomarker levels will be evaluated. Nailfold capillaroscopy parameters, including capillary density score and semi-quantitative morphological scores (tortuosity, dilatation, dystrophic changes, avascular areas, microhemorrhages, and neoangiogenesis), assessed using standardized nailfold capillaroscopy evaluation criteria, will be correlated with serum concentrations of asymmetric dimethylarginine (ADMA), von Willebrand factor (vWF), high-sensitivity C-reactive protein (hs-CRP), and D-dimer measured by laboratory assays. Correlation analysis will be performed to assess the relationship between microvascular structural alterations and biochemical markers of endothelial dysfunction, inflammation, and prothrombotic activity.
Correlation Between Occupational Radiation Exposure and Microvascular and Serum Biomarker Measurements | Baseline (cross-sectional analysis)
  The correlation between occupational radiation exposure and microvascular and biochemical parameters will be evaluated. Occupational radiation exposure will be assessed using self-reported work history, including duration of employment in radiation-related medical departments (years of exposure). Microvascular changes will be assessed by nailfold capillaroscopy using standardized semi-quantitative scoring systems, including capillary density score and morphological scores (tortuosity, dilatation, dystrophic changes, avascular areas, microhemorrhages, and neoangiogenesis). Biochemical parameters will include serum concentrations of asymmetric dimethylarginine (ADMA), von Willebrand factor (vWF), high-sensitivity C-reactive protein (hs-CRP), and D-dimer, measured by laboratory assays. Correlation analyses will be performed to evaluate the relationship between occupational radiation exposure duration and microvascular or serum biomarker measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Banu Yildiran, MD, Principal Investigator — Istanbul Training and Research Hospital, Dept. of Dermatology; Duygu Yamen, MD, Study Director — Istanbul Training and Research Hospital, Dept. of Dermatology; Ayse Esra Koku Aksu, MD, Prof, Study Chair — Istanbul Training and Research Hospital, Dept. of Dermatology
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes